CLINICAL TRIAL: NCT02219269
Title: A Complex Contraception Registry - UC Family Planning Collaborative Study
Brief Title: A Complex Contraception Registry
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other); University of California, San Francisco (Other); University of California, Irvine (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Sheila Mody, Assistant Professor, University of California, San Diego
Other Study IDs: 140166
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Diabetes; Cardiovascular Disease; Epilepsy; Migraine; Neurological Disorders; Cancer; Bariatric Surgery Candidate; Organ or Tissue Transplant; Complications; Lupus Erythematosus, Systemic; Other Hematologic Conditions; Other Venous Embolism and Thrombosis
Keywords: contraception; family planning; complex medical conditions
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Epilepsy; Migraine Disorders; Nervous System Diseases; Neoplasms; Lupus Erythematosus, Systemic; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Medically complex contraception users: Cohort includes women of reproductive age with diverse medical conditions (listed in inclusion criteria) who are referred to Family Planning felowship-trained physicians, seeking contraception counseling and administration.

SUMMARY:
The investigators will conduct a prospective observational cohort study to investigate factors that influence contraceptive method utilization among women with medical conditions. The investigators will also investigate how women with medical conditions access to contraception and family planning fellowship trained specialist. After the baseline questionnaire, there be a 3 month and 6 month follow up questionnaire to investigate continuation and satisfaction with the contraceptive method. This study is unique because it will allow us to explore doing collaborative family planning research at the multiple UC medical campuses.

DETAILED DESCRIPTION:
Many women with complex medical conditions who do not desire pregnancy do not receive contraception counseling from their primary or subspecialty care clinicians, and often they are not using contraception. This is an important deficiency as many have conditions that could worsen with pregnancy or for whom pregnancy can be complicated by the medical condition. Thus it is important for women with chronic disease to only become pregnant if they intend to do so. The United States Medical Eligibility Criteria for Contraceptive Use (USMEC), released in 2010, has greatly enhanced the ability of clinicians to counsel patient with complex medical conditions about their contraceptive options. It summarizes the safety of specific contraceptives when used on women with medical conditions. However, little is known about the contraceptive care of these women. We do not know if the availability of the USMEC has translated into evidence-based contraceptive counseling for these women. Further, little is known about their understanding of the interaction between their disease and pregnancy, their past experience and knowledge about contraception, and their contraceptive decision-making, satisfaction and continuation.

The purpose of the Complex Contraception Registry to is to recruit a cohort of women with complex medical conditions who are seen in contraception referral practices run by family planning fellowship trained physicians. We will assess their past experiences and baseline knowledge, their post-counseling experiences and choice of contraception, and their long-term satisfaction with and continuation of contraception. A multi-center registry is necessary because individual institutions see relatively few women with rare diseases such as a history of transplant surgery. The UC Family Planning Collaborative will facilitate recruitment of participants from the 5 UC medical campuses and will oversee their follow-up for one year.

Specific Aim include (1.) To investigate what factors influence contraceptive method utilization among women with complex medical conditions and their perceived risk of unintended pregnancy (2) To investigate how women with complex medical conditions access family planning fellowship trained specialist for contraception counseling and (3.) To assess satisfaction and continuation of contraceptive methods among women with complex medical conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Background: No limitation, will include minorities
2. Sexually Active with men
3. Diagnosis with at least one of the following conditions

   * Diabetes and other endocrine disorders
   * Cardiovascular Disease, such as Ischemic Heart Disease, Valvular disease, hypertension or pulmonary hypertension
   * Epilepsy, Migraine, and other neurologic disorders
   * History of or current cancer
   * History of or planning Bariatric Surgery
   * History of or planning Solid Organ Transplant
   * Systematic Lupus Erythematous and other rheumatologic conditions
   * History of or current Venous Thrombosis Embolism
   * Other Medical Conditions (such as Sickle Cell Disease or Cystic Fibrosis)

Exclusion Criteria:

1. Pregnant at time of recruitment
2. History of hysterectomy, bilateral oophorectomy, or sterilization procedure
3. Unable to provide informed consent
4. Attempting to become pregnant at time of recruitment
5. Not sexually active with men
6. No active telephone number or email for follow up

Women who are pregnant will be excluded from this study. However, no pregnancy testing will be conducted; pregnancy status will be based on self-reporting by subjects.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of women 18-45 years old and seeking contraception with the medical condition listed in inclusion criteria. Participants will be recruited from obstetrics and gynecology clinic at UCSD, UCLA, UCSF, UC Irvine and UC Davis. 250 participants will be enrolled. Approximately 50 cases will be recruited at each site.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Contraceptive method continuation and satisfaction | 6 month
  Questionnaire is used to report continued use and satisfaction with multiple choice answer: very satisfied, somewhat satisfied, dissatisfied. Questionnaires will be administered at 3 months and 6 months after recruitment.

SECONDARY OUTCOMES:
History of unintended pregnancy | 6 months
  Measured with questionnaire at baseline, 3 months, and 6 months
Change in Medical Condition | 6 months
  Measured with questionnaire at 3 months and 6 months
History of contraceptive methods used | 6 months
  Measured with questionnaire at baseline
If Contraception is Accessed in post-partum or post-abortion setting | 6 months
  Measured with questionnaire at baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jody Steinauer, MD, Principal Investigator — University of California, San Francisco; Radhika Rible, MD MS, Principal Investigator — University of California, Los Angeles; Tabetha Harken, MD MPH, Principal Investigator — UC Irvine; Catherine Cansino, MD MPH, Principal Investigator — UC Davis; Sheila Mody, MD MPH, Principal Investigator — UCSD
Locations (5):
- United States (5):
  - UCLA, Los Angeles, California
  - UC Irvine, Orange, California
  - UC Davis, Sacramento, California
  - UCSD, San Diego, California
  - UCSF, San Francisco, California

REFERENCES:
- [Background] Center for Disease Control and Prevention. U.S Medical Eligibility Criteria for Contraceptive Use, 2010.MMWR 2010;59 (No.RR-4).76-81
- [Derived] Mody SK, Cansino C, Rible R, Farala JP, Steinauer J, Harken T; University of California Family Planning Collaborative. Contraceptive use among women with medical conditions: Factors that influence method choice. Semin Perinatol. 2020 Aug;44(5):151310. doi: 10.1016/j.semperi.2020.151310. Epub 2020 Aug 20. PMID 32888723